CLINICAL TRIAL: NCT00001084
Title: A Prospective Randomized Double-Blind Trial of Three Maintenance Regimens for HIV-Infected Subjects Receiving Induction Therapy With Zidovudine, Lamivudine and Indinavir
Brief Title: A Study of Three Treatment Combinations Using Zidovudine Plus Lamivudine Plus Indinavir in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 343; 11314 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Prospective Studies; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Indinavir; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To compare the proportion of patients who sustain suppression of plasma HIV RNA to undetectable levels [AS PER AMENDMENT 09/19/97: below 200 copies/mL by Roche UltraSensitive assay] among the 3 regimens during the maintenance phase.

The objective of antiretroviral therapy is to reduce HIV replication, preserve immunologic function and delay the development of HIV-related complications. In patients administered potent antiretroviral regimens, HIV RNA levels are reduced below 500 copies/ml of plasma and below the level of detection of commercially available assays. This protocol attempts to learn if a less intensive regimen can successfully sustain viral suppression after induction with a triple-drug regimen. The study also addresses whether HIV can be eradicated in patients following prolonged treatment with induction and maintenance regimens.

DETAILED DESCRIPTION:
The objective of antiretroviral therapy is to reduce HIV replication, preserve immunologic function and delay the development of HIV-related complications. In patients administered potent antiretroviral regimens, HIV RNA levels are reduced below 500 copies/ml of plasma and below the level of detection of commercially available assays. This protocol attempts to learn if a less intensive regimen can successfully sustain viral suppression after induction with a triple-drug regimen. The study also addresses whether HIV can be eradicated in patients following prolonged treatment with induction and maintenance regimens.

All patients will receive open label induction therapy with zidovudine (ZDV), lamivudine (3TC) and indinavir (IDV) for 6 months. Following the 6 month induction phase, patients with undetectable plasma HIV RNA at weeks 16, 20 and 24 will enter the maintenance phase [blinded maintenance phase AS PER AMENDMENT 09/19/97] and be randomized to one of three maintenance regimens, i.e., either continued ZDV/3TC/IDV (control), or ZDV/3TC/IDV placebo or ZDV placebo/3TC placebo/IDV. Prior to randomization, patients are stratified according to entry HIV RNA level (greater than or equal to 30,000 or less than 30,000 copies/ml) and by prior ZDV therapy (at least 7 days or less than 7 days). After 12 months [AS PER AMENDMENT 09/19/97: 18 months] of maintenance therapy, treatment will be withdrawn at 6-month intervals in randomly-selected patients who have achieved undetectable HIV RNA. AS PER 09/19/97 AMENDMENT: After 18 months of blinded maintenance therapy, treatment is unblinded for patients whose HIV RNA levels remain detectable. Such patients receive optimal therapy, either continuing the protocol regimen or initiating alternative therapy.

AS PER AMENDMENT 2/27/98: An interim review conducted in January, 1998 demonstrated that the strategy of less intensive antiviral therapy after 6 months of IDV/3TC/ZDV induction therapy is less effective than continuation of triple drug therapy except for ZDV-naive patients assigned to ZDV/3TC. Therefore, the maintenance phase of this study has been discontinued.

Patients currently on blinded maintenance are unblinded immediately and have the option of reinitiating open-label triple therapy with IDV/3TC/ZDV or discontinuing study treatment. Patients currently on induction may register for continued open-label triple therapy or may discontinue study treatment. This amendment allows treatment extension so that subjects may receive open-label triple therapy until May 31, 1998. At that time, a rollover protocol or another modification with a longer period of drug supply may become available. Patients who choose to go off treatment are followed until May 31, 1998.

AS PER AMENDMENT 04/23/98: This study will now provide treatment with open-label ZDV/3TC/IDV until August 1, 1998. A rollover protocol or another 343 protocol modification with a longer period of drug supply may become available, but this cannot be guaranteed.

AS PER AMENDMENT 06/19/98: This study will now provide treatment with open-label ZDV/3TC/IDV until either November 1, 1998 or until 3 months after the rollover study (A5025) is available to the study sites (whichever comes first).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* A CD4 cell count >= 200 cells/mm3 within 90 days prior to study entry.
* Plasma HIV RNA >= 1000 copies/ml within 90 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following conditions or symptoms are excluded:

* A malignancy that requires systemic chemotherapy.

Concurrent Medication:

Excluded:

* Oral ketoconazole (Nizoral), terfenadine (Seldane), astemizole (Hismanal), cisapride (Propulsid), triazolam (Halcion) or midazolam (Versed).
* All antiretroviral therapies other than study medications.
* Rifabutin and rifampin.
* Investigational drugs and vaccines.
* Systemic cytotoxic chemotherapy.
* Interferon, interleukins, GM-CSF and HIV vaccines.

Patients with any of the following prior conditions are excluded:

* Unexplained temperature > 38.5 degrees C for any 7 days within 30 days prior to study entry.
* Chronic diarrhea as defined as > 3 liquid stools per day persisting for 15 days within 30 days prior to study entry.
* Proven or suspected acute hepatitis within 30 days prior to study entry, even if AST and ALT are <= 5.0 X ULN (upper limit of normal).
* A history of >= Grade 2 bilateral peripheral neuropathy within 60 days prior to study entry.
* A history of intolerance to 300 mg/day of ZDV defined as any toxicity requiring a dose reduction or termination of ZDV.

Prior Medication:

Excluded:

* Acute therapy for an infection or other medical illness within 14 days prior to study entry.
* Any prior therapy with 3TC or experimental drug 1592.
* More than 2 weeks of lifetime exposure to protease inhibitor therapy; any exposure within 14 days prior to study entry.
* Interferons, interleukins, GM-CSF or HIV vaccines within 30 days prior to study entry.
* Any experimental therapy (drugs or vaccines) within 30 days prior to study entry.
* Rifampin or rifabutin within 14 days prior to study entry.
* Systemic cytotoxic chemotherapy within 30 days prior to study entry.
* Oral ketoconazole (Nizoral), terfenadine (Seldane), astemizole (Hismanal), cisapride (Propulsid), triazolam (Halcion) or midazolam (Versed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Study Completion 1997-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Havlir D, Study Chair; Richman D, Study Chair
Locations (45):
- United States (45):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Tulane Med Ctr Hosp, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Havlir DV, Marschner IC, Hirsch MS, Collier AC, Tebas P, Bassett RL, Ioannidis JP, Holohan MK, Leavitt R, Boone G, Richman DD. Maintenance antiretroviral therapies in HIV-infected subjects with undetectable plasma HIV RNA after triple-drug therapy. AIDS Clinical Trials Group Study 343 Team. N Engl J Med. 1998 Oct 29;339(18):1261-8. doi: 10.1056/NEJM199810293391801. PMID 9791141
- [Background] Bowersox J. ACTG 343: three drugs better than two for maintaining HIV suppression. NIAID AIDS Agenda. 1998 Mar:1-2, 10-1. PMID 11365088
- [Background] Maenza JR. ACTG 343: (why) we can't relax our grip on viral suppression. Hopkins HIV Rep. 1998 May;10(3):10. PMID 11365491
- [Background] O'Brien TR, McDermott DH, Ioannidis JP, Carrington M, Murphy PM, Havlir DV, Richman DD. Effect of chemokine receptor gene polymorphisms on the response to potent antiretroviral therapy. AIDS. 2000 May 5;14(7):821-6. doi: 10.1097/00002030-200005050-00008. PMID 10839590
- [Background] Zhou XJ, Havlir DV, Richman DD, Acosta EP, Hirsch M, Collier AC, Tebas P, Sommadossi JP; AIDS Clinical Trials Study 343 Investigators. Plasma population pharmacokinetics and penetration into cerebrospinal fluid of indinavir in combination with zidovudine and lamivudine in HIV-1-infected patients. AIDS. 2000 Dec 22;14(18):2869-76. doi: 10.1097/00002030-200012220-00008. PMID 11153668
- [Background] Havlir DV, Bassett R, Levitan D, Gilbert P, Tebas P, Collier AC, Hirsch MS, Ignacio C, Condra J, Gunthard HF, Richman DD, Wong JK. Prevalence and predictive value of intermittent viremia with combination hiv therapy. JAMA. 2001 Jul 11;286(2):171-9. doi: 10.1001/jama.286.2.171. PMID 11448280
- [Background] Seth A, Markee J, Ap S, Sevin A, Hoering A, Hirsch M, Collier A, Letvin N, McElrath MJ. Alterations in T cell phenotype and antigen-specific cytotoxicity in patients receiving three anti-retroviral agents (ACTG protocol 343). Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:132 (abstract no 340)
- [Background] Havlir DV, Hirsch M, Collier A, Marschner I, Bassett R, Tebas P, Ioannidis J, Richman DD. Randomized trial of indinavir (IDV) vs. zidovudine (ZDV)/lamivudine (3TC) vs IDV/ZDV/3TC maintenance therapy after induction IDV/ZDV/3TC therapy. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:225 (abstract no LB16)
- [Background] Gunthard HF, Havlir DV, Fiscus S, Zhang ZQ, Eron J, Mellors J, Gulick R, Frost SD, Brown AJ, Schleif W, Valentine F, Jonas L, Meibohm A, Ignacio CC, Isaacs R, Gamagami R, Emini E, Haase A, Richman DD, Wong JK. Residual human immunodeficiency virus (HIV) Type 1 RNA and DNA in lymph nodes and HIV RNA in genital secretions and in cerebrospinal fluid after suppression of viremia for 2 years. J Infect Dis. 2001 May 1;183(9):1318-27. doi: 10.1086/319864. Epub 2001 Apr 10. PMID 11294662
- [Background] Gulick RM, Mellors J, Havlir D, Eron J, Gonzalez C, McMahon D, Richman D, Valentine F, Rooney J, Jonas L, Meibohm A, Emini E, Chodakewitz J. Potent and sustained antiretroviral activity of indinavir (IDV), zidovudine (ZDV) and lamivudine (3TC). Int Conf AIDS. 1996 Jul 7-12;11(Program Supplement):19 (abstract no ThB931)